CLINICAL TRIAL: NCT04552483
Title: Effects of Nitazoxanide Administration to Patients in the Initial Phase of COVID-19
Brief Title: Effects of Early Use of Nitazoxanide in Patients With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Ministry of Science and Technology, Brazil (Other); National Research Council, Brazil (Other); ATCGen (Unknown); Complexo Hospitalar Municipal de São Caetano do Sul (Unknown); Hospital de Transplante Doutor Euryclides de Jesus Zerbini (Other); Secretaria Municipal de Saúde de Bauru (Unknown); Santa Casa de Misericórdia de Sorocaba (Unknown); Secretaria Municipal de Saúde de Guarulhos (Unknown); Hospital e Maternidade Therezinha de Jesus (Unknown); Secretaria de Estado de Saúde do Distrito Federal (Unknown)
Responsible Party: Principal Investigator, Jose Roberto Lapa e Silva, Clinical Investigator, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SARITA-2; RBR-4nr86m (Other: Registro Brasileiro de Ensaios Clínicos (REBEC)); 32258920.0.1001.5257 (Other: Comitê Nacional de Ética em Pesquisa (CONEP))
Record Dates: First submitted 2020-09-09; First posted 2020-09-17 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Covid19; Coronavirus
Keywords: covid19; coronavirus; early treatment; COVID-19; new coronavirus; treatment; brazil; nitazoxanide
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — nitazoxanide

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with COVID-19 will be randomly divided into 2 groups: experimental and control groups.
  Experimental group: 196 patients diagnosed with COVID-19 confirmed by RT-PCR will receive nitazoxanide 500mg 8/8 hs for 5 days. Control group: 196 patients diagnosed with COVID-19 confirmed by RT-PCR will receive placebo 8/8 hs for 5 days.
Who Masked: Participant, Care Provider
Masking Description: Patients were randomly allocated into one of the two groups: A or B. Patients received labelled medication: A or B, by the pharmacist. Patients received an identification number, so care providers, outcomes assessors and investigators did not know anything regarding the patients' groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitazoxanide (Experimental): Patients received nitazoxanide 500mg 8/8hours, for 5 days.
  Interventions: Drug: Nitazoxanide
- Placebo (Placebo Comparator): Patients received placebo 500mg 8/8hours, for 5 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitazoxanide — Nitazoxanide 500mg 8/8 hours for 5 days in the early clinical phase of COVID-19.
  Other Names: azox; annita; irose; tanisea; trinida; zoxany
  Arms: Nitazoxanide
Drug: Placebo — Placebo 8/8 hours for 5 days in the early clinical phase of COVID-19.
  Arms: Placebo

SUMMARY:
Multicenter, randomized, placebo-controlled, parallel, blinded, interventional, treatment clinical trial with two arms.

Population: 392 Patients with COVID-19 (Coronavirus Disease-19), confirmed by RT-PCR (Real Time polymerase chain reaction), symptomatic in the early phase of the disease.

Experimental group: 196 patients, nitazoxanide 500mg 8 / 8 hours for 5 days. Control group: 196 patients, placebo 8/8 hours for 5 days.

DETAILED DESCRIPTION:
SARITA-2 is a multicenter, randomized, placebo-controlled, parallel, -blinded, interventional, treatment clinical trial with two arms, which aims to study the impact of nitazoxanide in the early phase of the COVID-19 (Coronavirus Disease-19).

Experimental group: 196 patients received nitazoxanide 500mg 8 / 8 hours for 5 days. Control group: 196 patients received placebo 8/8 hours for 5 days.

Population: 392 Patients with COVID-19, confirmed by RT-PCR (Real Time polymerase chain reaction), symptomatic in the early phase of the disease.

Calculation of the sample size was based on a previous study which demonstrated that 78% of Covid-19 patients in group 4 (Hospitalized without oxygen therapy), according to the WHO ordinal classification, experienced complete resolution of symptoms after receiving placebo.10 In the present trial, patients were classified as group 2 (Symptomatic and independent), and a greater degree of recovery as measured by symptom-free days (80%) was expected even after placebo. Thus, assuming an 11% increase in symptom-free days in those patients who would receive nitazoxanide compared to placebo, we would need approximately 196 patients per experimental group, admitting a beta error of 15% and alpha error of 5%, for a total n of 392 patients. Calculation of the sample size was done by G*Power 3.1.9.2 (Universität Düsseldorf, Düsseldorf, Germany).

ELIGIBILITY:
Inclusion Criteria:

* Clinical scenario compatible with infection by the SARS-CoV-2 [Characteristic symptoms of COVID-19 (fever and / or cough and / or fatigue)
* Beginning 1 to 3 days before inclusion in the study
* Age equal or superior to 18 years
* Willingness to receive study treatment
* Providing written and informed consent or the same consent signed by a family member

Exclusion Criteria:

* Negative result of RT-PCR for SARS-COV2 collected on admission
* Impossibility to use oral medications
* History of severe liver disease (Child Pugh C class)
* Previous renal failure
* Severe heart failure (NYHA 3 or 4)
* COPD (GOLD 3 and 4)
* Neoplasia in the last 5 years
* Known autoimmune disease
* Individuals with known hypersensitivity to study drug
* Previous treatment with the study medication during the last 30 days
* Clinical suspicion of tuberculosis and bacterial pneumonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-09-05 (Actual)

PRIMARY OUTCOMES:
Days with fever | Day8
  Reduction in the duration of fever of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide compared to patients treated with placebo; verified through the collection of information with the patient; quantified by the number of days that presented the symptom.
Days with cough | Day8
  Reduction in the duration of cough of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide compared to patients treated with placebo; verified through the collection of information with the patient; quantified by the number of days that presented the symptom.
Days with asthenia | Day8
  Reduction in the duration of asthenia of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide compared to patients treated with placebo; verified through the collection of information with the patient; quantified by the number of days that presented the symptom.

SECONDARY OUTCOMES:
SARS-COV-2 viral load - absolute number | Day1
  Compare the evolution of viral load in naso- and oropharyngeal swab in patients with COVID-19 treated with nitazoxanide or placebo on day 1; verified using the RT-PCR technique; quantified by the absolute number
SARS-COV-2 viral load - absolute number | Day8
  Compare the evolution of viral load in naso- and oropharyngeal swab in patients with COVID-19 treated with nitazoxanide or placebo on day 8; verified using the RT-PCR technique; quantified by the absolute number.
SARS-COV-2 viral load - percentage | Day 1
  Compare the evolution of viral load in naso- and oropharyngeal swab in patients with COVID-19 treated with nitazoxanide or placebo on day 1; verified using the RT-PCR technique; quantified by the percentage change between the two groups.
SARS-COV-2 viral load - percentage | Day 8
  Compare the evolution of viral load in naso- and oropharyngeal swab in patients with COVID-19 treated with nitazoxanide or placebo on day 8; verified using the RT-PCR technique; quantified by the percentage change between the two groups.
Hospital admission rate - absolute number | Day8
  Compare the hospital admission rate of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, in the period of 8 days; verified by information actively collected from patients or family members; quantified by absolute number.
Hospital admission rate - percentage | Day8
  Compare the hospital admission rate of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, in the period of 8 days; verified by information actively collected from patients or family members; quantified by percentage.
Serum Interleukin-6 | Day 3
  Compare the levels of inflammatory mediators: (interleukin [IL] -6 from patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 3; verified by the measurement of cytokines in patient serum by the ELISA technique; quantified by the absolute number between the two groups.
Serum Interleukin-6 | Day 8
  Compare the levels of inflammatory mediators: (interleukin [IL] -6 from patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 8; verified by the measurement of cytokines in patient serum by the ELISA technique; quantified by the absolute number between the two groups.
Serum Interleukin-1-beta | Day 3
  Compare the levels of inflammatory mediators: IL-1-beta from patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 3; verified by the measurement of cytokines in patient serum by the ELISA technique; quantified by the absolute number between the two groups.
Serum Interleukin-1-beta | Day 8
  Compare the levels of inflammatory mediators: IL-1-beta from patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 8; verified by the measurement of cytokines in patient serum by the ELISA technique; quantified by the absolute number between the two groups.
Serum Interleukin-8 | Day 3
  Compare the levels of inflammatory mediators: IL-8 from patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 3; verified by the measurement of cytokines in patient serum by the ELISA technique; quantified by the absolute number between the two groups.
Serum Interleukin-8 | Day 8
  Compare the levels of inflammatory mediators: IL-8 from patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 8; verified by the measurement of cytokines in patient serum by the ELISA technique; quantified by the absolute number between the two groups.
Serum tumor necrosis factor (TNF)-alfa | Day 3
  Compare the levels of inflammatory mediators: tumor necrosis factor (TNF)-alfa from patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 3; verified by the measurement of cytokines in patient serum by the ELISA technique; quantified by the absolute number between the two groups.
Serum tumor necrosis factor (TNF)-alfa | Day 8
  Compare the levels of inflammatory mediators: tumor necrosis factor (TNF)-alfa from patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 8; verified by the measurement of cytokines in patient serum by the ELISA technique; quantified by the absolute number between the two groups.
Serum interferon-gamma | Day 3
  Compare the levels of inflammatory mediators: interferon-gamma from patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 3; verified by the measurement of cytokines in patient serum by the ELISA technique; quantified by the absolute number between the two groups.
Serum interferon-gamma | Day 8
  Compare the levels of inflammatory mediators: interferon-gamma from patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 8; verified by the measurement of cytokines in patient serum by the ELISA technique; quantified by the absolute number between the two groups.
Serum monocyte chemoattractant protein (MCP)-1 | Day 3
  Compare the levels of inflammatory mediators: monocyte chemoattractant protein (MCP)-1 from patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 3; verified by the measurement of cytokines in patient serum by the ELISA technique; quantified by the absolute number between the two groups.
Serum monocyte chemoattractant protein (MCP)-1 | Day 8
  Compare the levels of inflammatory mediators: monocyte chemoattractant protein (MCP)-1 from patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 8; verified by the measurement of cytokines in patient serum by the ELISA technique; quantified by the absolute number between the two groups.
Complete blood count | Day 3
  Evaluate evolution of complete blood count with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 3; verified by laboratory tests and expressed by the absolute number between the two groups.
Complete blood count | Day 8
  Evaluate evolution of complete blood count with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 8; verified by laboratory tests and expressed by the absolute number between the two groups.
C-reactive protein - absolute number | Day 3
  To evaluate the levels of C-reactive protein (CRP) of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 3; verified by laboratory tests and expressed by the absolute number between the two groups.
C-reactive protein - absolute number | Day 8
  To evaluate the levels of C-reactive protein (CRP) of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 8; verified by laboratory tests and expressed by the absolute number between the two groups.
C-reactive protein - percentage | Day 3
  To evaluate the levels of C-reactive protein (CRP) of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 3; verified by laboratory tests and expressed by the percentage between the two group.
C-reactive protein - percentage | Day 8
  To evaluate the levels of C-reactive protein (CRP) of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 8; verified by laboratory tests and expressed by the percentage between the two groups.

OTHER OUTCOMES:
Adverse events - percentage | Day 8
  Assess the incidence and profile of adverse events reported throughout the study, by treatment group; verified by information actively collected from patients or family members; quantified by percentage.
Adverse events - absolute number | Day8
  Assess the incidence and profile of adverse events reported throughout the study, by treatment group; verified by information actively collected from patients or family members; quantified by absolute number.
Treatment discontinuation rate - absolute number | Day8
  Assess the rate of treatment discontinuation due to adverse events; verified by information actively collected from patients or family members; quantified by absolute number.
Treatment discontinuation rate - percentage | Day8
  Assess the rate of treatment discontinuation due to adverse events; verified by information actively collected from patients or family members; quantified by percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia RM Rocco, MD, PhD, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Universidade Federal do Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan on sharing all IPD that underlie results in a publication for editorial board, with cautious of not sharing confidential data.
Supporting Information: Study Protocol
Time Frame: Available as soon as the editorial board of the journal accepting the manuscript requires.
Access Criteria: Editorial board of the Journal accepting the manuscript.

REFERENCES:
- [Background] Rossignol JF. Nitazoxanide, a new drug candidate for the treatment of Middle East respiratory syndrome coronavirus. J Infect Public Health. 2016 May-Jun;9(3):227-30. doi: 10.1016/j.jiph.2016.04.001. Epub 2016 Apr 16. PMID 27095301
- [Background] Rossignol JF. Nitazoxanide: a first-in-class broad-spectrum antiviral agent. Antiviral Res. 2014 Oct;110:94-103. doi: 10.1016/j.antiviral.2014.07.014. Epub 2014 Aug 7. PMID 25108173
- [Background] Rajoli RK, Pertinez H, Arshad U, Box H, Tatham L, Curley P, Neary M, Sharp J, Liptrott NJ, Valentijn A, David C, Rannard SP, Aljayyoussi G, Pennington SH, Hill A, Boffito M, Ward SA, Khoo SH, Bray PG, O'Neill PM, Hong WD, Biagini G, Owen A. Dose prediction for repurposing nitazoxanide in SARS-CoV-2 treatment or chemoprophylaxis. medRxiv [Preprint]. 2020 May 6:2020.05.01.20087130. doi: 10.1101/2020.05.01.20087130. PMID 32511548
- [Background] Pepperrell T, Pilkington V, Owen A, Wang J, Hill AM. Review of safety and minimum pricing of nitazoxanide for potential treatment of COVID-19. J Virus Erad. 2020 Apr 30;6(2):52-60. doi: 10.1016/S2055-6640(20)30017-0. PMID 32405422